CLINICAL TRIAL: NCT05795816
Title: The Effectiveness of Testofen on Energy, Fatigue, Mental Acuity, and Other Quality of Life Symptoms Post COVID-19 Infection
Brief Title: Effectiveness of Testofen Compared to Placebo on Long COVID Symptoms
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: RDC Clinical Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FENCOV
Record Dates: First submitted 2023-03-27; First posted 2023-04-03 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2024-10

CONDITIONS: Long Covid19
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Testofen (Active Comparator): Testofen in capsule form - taken as 2 x 300 mg daily with food (1 in the morning and 1 in the evening)
  Interventions: Drug: Testofen
- Microcrystalline cellulose (Placebo Comparator): Microcrystalline cellulose in capsule form - taken as per Active comparator
  Interventions: Drug: Microcrystalline cellulose

INTERVENTIONS:
Drug: Testofen — Twice daily dose of 1 capsule (300mg per capsule Testofen)
  Arms: Testofen
Drug: Microcrystalline cellulose — Twice daily dose of 1 capsule
  Arms: Microcrystalline cellulose

SUMMARY:
This is a double blind, randomised, placebo-controlled trial to evaluate orally-dosed Testofen (a specialised extract of Trigonella foenum-graecum (Fenugreek) seed) compared to placebo on post COVID-19 symptoms in otherwise healthy participants 18 years and over.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years and over
* Able to provide informed consent
* Diagnosed with COVID-19 infection (RAT or PCR test) >4 weeks, but < 12 months and experiencing post COVID symptoms (1)
* Agree not to participate in another clinical trial while enrolled in this trial

  1. Common post COVID symptoms may include fatigue, cough, chest pain, hair loss, weakness, joint pain, cardiac issues, neurocognitive impairment including memory loss, and decreased quality of life

Exclusion Criteria:

* Symptoms resulting from vaccination (2)
* Unstable or serious illness (e.g., serious mood disorders, neurological disorders such as MS, kidney disease, liver disease, heart conditions, diabetes, thyroid gland dysfunction) (3)
* Current malignancy (excluding BCC) or chemotherapy and radiotherapy treatment for malignancy within the previous 2 years
* Receiving/prescribed coumandin (Warfarin), heparin, dalteaparin, enoxaparin or other anticoagulation therapy
* Receiving pharmaceutical treatment for anxiety, libido, low energy
* Active smokers, nicotine use, alcohol, or drug (prescription or illegal substances) abuse
* Chronic past and/or current alcohol use (>14 alcoholic drinks per week)
* Allergic to any of the ingredients in the active or placebo formula
* Known pregnant or lactating women
* Any condition which in the opinion of the investigator makes the participant unsuitable for inclusion
* Participants who have participated in any other related clinical study during the past 1 month
* History of infection in the month prior to the study

  (2) Symptoms must be as a direct result of having contracted COVID. If symptoms only appeared within 2 weeks of a vaccination it will be considered a vaccine injury and not classed as a result of COVID.

  (3) An unstable illness is any illness that is currently not being treated with a stable dose of medication or is fluctuating in severity. A serious illness is a condition that carries a risk of mortality, negatively impacts quality of life and daily function and/or is burdensome in symptoms and/or treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2023-10-25 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Change in Energy and Fatigue | Baseline, week 4, week 8 and week 12
  Change in energy and fatigue as measured via Fatigue Severity Scale. The items are scored on a 7 point scale with 1 = strongly disagree and 7= strongly agree. The minimum score = 9 and maximum score possible = 63. Higher the score = greater fatigue severity
Change in Energy and Fatigue | Baseline, week 4, week 8 and week 12
  Change in energy and fatigue as measured via Global Fatigue Index. The items are scored on a 10 point scale with 1 = not at all and 10 = great deal. Higher he score = greater fatigue

SECONDARY OUTCOMES:
Change in Memory | Baseline, week 4, week 8 and week 12
  Change in Memory as measured by Short Term Memory testing
Change in Mental Acuity | Baseline, week 4, week 8 and week 12
  Change in Mental acuity as measured by Reaction Time Test
Change in Muscle Strength (Hand grip) | Baseline, week 4, week 8 and week 12
  Change in Muscle Strength (Hand grip) as measured by Dynamometer
Change in Hair loss/growth | Baseline, week 4, week 8 and week 12
  Change in Hair loss/growth as measured by Hair loss questionnaire
Change in Libido | Baseline, week 4, week 8 and week 12
  Change in Libido as measured by - If male, DISF-SR (Derogatis Sexual Function Index), If female, FSFI (Female Sexual Function Index)
Change in Stress and Mood | Baseline, week 4, week 8 and week 12
  Change in Stress and Mood via Depression Anxiety and Stress Scale (DASS-21)
Change in Quality of Life Indicators | Baseline, week 4, week 8 and week 12
  Change in Quality of Life Indicators via Symptom Burden Questionnaire - Long Covid
Change in Pathology results via Blood test | Baseline, week 4, week 8 and week 12
  Change in Pathology results (Full blood count, CRP, iron, Soluble P-selectin, Testosterone, DHT, SHBG, Estrogen, IGF1, Cortisol, Prostaglandins, Inflammatory markers IL-10, IL-6, IL-17, TNF-a) as measured by Blood test
Change in Weight | Baseline, week 4, week 8 and week 12
  Change in Weight as measured by scales in kg
Height | Baseline, week 4, week 8 and week 12
  Height as measured by tape measure in centimetres
Change in Safety as assessed by Adverse Events Recording | During enrolment period
  Change in Safety as assessed by Adverse Events Recording
Change in safety markers as assessed by pathology | Baseline, week 4, week 8 and week 12
  Change in safety markers E/LFT as assessed by pathology

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Rao, PhD, Principal Investigator — RDC Clinical Pty Ltd
Locations (1):
- RDC Clinical Pty Ltd, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared